CLINICAL TRIAL: NCT05545436
Title: A Single-center Prospective Single-arm Study of the Efficacy of Carrelizumab (PD-1) Combined With Chemotherapy in Neoadjuvant Treatment of Locally Advanced Gastric Cancer and Its Effect on Tumor Immune Microenvironment
Brief Title: Carrelizumab (PD-1) Combined With Chemotherapy in Neoadjuvant Treatment of Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hongbo Wei, The director of Gastrointestinal Surgery, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: （2022）02-181-01
Record Dates: First submitted 2022-09-13; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — camrelizumab; Oxaliplatin; XELOX; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + SOX (oxaliplatin + Teggio) /XELOX (oxaliplatin + capecitabine ) (Experimental): Camrelizumab + SOX / XELOX
  Interventions: Drug: Camrelizumab + SOX (oxaliplatin + Teggio) /XELOX (oxaliplatin + capecitabine )

INTERVENTIONS:
Drug: Camrelizumab + SOX (oxaliplatin + Teggio) /XELOX (oxaliplatin + capecitabine ) — Camrelizumab + SOX (oxaliplatin + Teggio) /XELOX (oxaliplatin + capecitabine ) Drug: Camrelizumab 200mg Drug: oxaliplatin 130 mg/m2 Drug: Teggio 40 mg/m2 Drug: oxaliplatin 130 mg/m2 Drug: capecitabine 1000 mg/m2 Q3W for 3 cycles. Radical surgery was performed 3 weeks after the last neoadjuvant treatment.
  Other Names: Camrelizumab + SOX / XELOX

SUMMARY:
This is a single-arm, open, exploratory clinical study to evaluate the efficacy of carrelizumab (PD-1) combined with chemotherapy (SOX/XELOX) as neoadjuvant therapy and to observe the changes of tumor immune microenvironment in patients with locally advanced gastric or gastroesophageal junction cancer (T3-4NXM0).

DETAILED DESCRIPTION:
For advanced gastric cancer, standard treatment is D2 gastrectomy combined with perioperative medications, when the tumor is infiltrating into submucosa, around or with lymph node metastasis, and can reduce the success rate of surgery, previous studies have showed a tumor on perioperative chemotherapy helps to drop period, and improve the long-term survival of patients, compared with surgery alone, It can improve the 5-year overall survival (OS) by about 10%. At present, SOX protocol is recommended as the perioperative protocol for advanced gastric cancer in domestic guidelines [5]. However, for patients with T3/T4 or positive lymph node (N+), the probability of recurrence or metastasis after resection is high, and the 5-year survival rate is only 23%. Previous studies have found that the prognosis of patients with complete pathological response or near complete pathological response after neoadjuvant chemotherapy is significantly improved, whereas the pCR rate is only less than 10%. It is an effective way to improve the prognosis of gastric cancer patients to seek neoadjuvant therapy that can improve the pathological response rate. Chemotherapy and immune checkpoint inhibitor drugs have a synergistic mechanism on the theoretical basis. Pd-1 inhibitors are a kind of immune checkpoint inhibitors. In the process of "immune escape" of tumors,PD-1 inhibitors are involved in the activation process of the immune system, and by inhibiting PD-1 receptors, T cells can be activated normally. Thus, the immune system of the body can promote the killing of tumor cells.

Our research group plans to carry out the study of carrelizumab (PD-1) combined with SOX/XELOX chemotherapy as a neoadjuvant therapy in locally advanced gastric cancer. A total of 34 patients with locally advanced gastric or gastroesophageal junction carcinoma of T3-4NXM0 were enrolled. After 3 cycles of carrelizumab (PD-1) combined with chemotherapy, radical resection was performed, and the treatment effect was evaluated by pathological remission of the surgical tissue. Collection and treatment of gastroscope biopsy tissue samples before and after neoadjuvant therapy surgery samples: 1. The multiple fluorescent immunohistochemical (mIHC) technique were used to detect the immune cells in tumor tissue infiltration, compared neoadjuvant therapy after curative effect before treatment between patients with good and poor effects of immune cell infiltration, the difference between a explore treatment response and the correlation between the baseline immune microenvironment; To compare the changes of immune cell infiltration before and after treatment, and to explore the effect of combined immunotherapy on the immune microenvironment of locally advanced gastric cancer. 2. High-throughput sequencing technology was used to sequence DNA molecules to compare the pre-treatment gene sequences between patients with good and poor efficacy after neoadjuvant therapy, and to explore the correlation between the effect of neoadjuvant therapy and gene sequence changes (dMMR, MSI, TMB, PD-L1, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. T3-4NxM0 locally advanced gastric or gastroesophageal junction carcinoma was confirmed by gastroscopic biopsy, CT and pathological examination;
2. No previous systematic treatment for the current disease;
3. Age ≥ 70 years, age ≥18 years, both sexes;
4. ECOG physical status score 0-1; Full organ and bone marrow function:
5. Blood routine: hemoglobin ≥90g/L, neutrophil count ≥1.5×10^9/L, platelet count ≥75×10^9/L; Liver function: serum total bilirubin ≤1.5× upper normal value (UNL), aspartate transferase ≤3×UNL, alanine Acid transferase ≤3×UNL; Renal function: serum creatinine ≤1.5×UNL, creatinine clearance rate ≥50ml/min; Coagulation function: INR, APTT and PT ≤1.5×UNL; Serum albumin ≥30g/L; Thyrotropin (TSH) and free thyroxine (fT4) were within the range of normal ±10%.

   Electrocardiogram showed no obvious abnormality.
6. Not receiving blood transfusion, blood products, or blood cell growth factors such as granulocyte colony-stimulating factor within 2 weeks;
7. Sign an informed consent form before starting the study on a specific screening procedure;
8. The estimated survival time is more than 3 months;
9. Subjects volunteered to join this study, with good compliance, safety and survival follow-up -

Exclusion Criteria:

Patients with any of the following were excluded from the study:

1. People with allergic disease, history of severe drug allergy, known allergy to macromolecular protein preparations or carrelizumab;
2. Early gastric cancer;
3. Gastric cancer patients with HER2 amplification by pathological gene detection;
4. History of other malignancies (except cured basal cell carcinoma of the skin, cured cervix) with disease-free survival <5 years Carcinoma in situ and gastrointestinal neoplasms proven to be cured by endoscopic mucosal resection);
5. The presence or history of any active autoimmune disease (including but not limited to: interstitial pneumonia, Uveitis, enteritis, nephritis, hyperthyroidism, hypothyroidism);
6. You are using immunosuppressive agents or hormone therapy (systemic or topical) to achieve immunosuppression, and Continued to use within 2 weeks before enrollment;
7. Severe infection (if intravenous antibiotics, antifungal or antiviral drugs are needed);
8. Congenital or acquired immune deficiency (such as HIV-infected persons), or active hepatitis ((with regular antiviral treatment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR, Becker criteria, TRG 1A) | Up to approximately 6 months.
  It was evaluated according to tumor regression grade (Becker standard) : TRG1a had no residual cancer; TRG1b < 10% residual cancer; TRG2 10%-50% residual cancer; TRG3 > 50% residual cancer.

SECONDARY OUTCOMES:
Major pathological response rate (MPR, TRG1a/ B) | Up to approximately 6 months.
  It was referred to Tumor Regression Grade (Becker Standard) as above.
R0 resection rate and objective response rate (ORR, RECIST 1.1) | Up to approximately 6 months.
  It was evaluated using the Response Assessment criteria for Solid tumors (RECIST 1.1). Subjects were required to have a measurable tumor lesion at baseline, and the outcome was classified as complete response (CR), partial response (PR), stable response (SD), and progressive response (PD) according to RECIST 1.1 criteria. Immune-related pseudoresults needed to be reconfirmed. During the screening period, baseline tumor imaging evaluation was completed within 4 weeks before the first treatment.Clinical tumor imaging evaluation was performed every 2 weeks during treatment. If disease progression was first reported according to RECIST 1.1, a clinical imaging confirmation was required 4 weeks later according to irRC. Investigators may add unplanned tumor imaging as clinically necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Wei, M.D., Ph.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China